CLINICAL TRIAL: NCT04454866
Title: Effects of Penehyclidine in Preventing Postoperative Nausea and Vomiting in Patients Underging Bimaxillary Surgery: A Randomised Controlled Trial
Brief Title: Penehyclidine for Prevention of Nausea and Vomiting After Bimaxillary Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Hospital of Stomatology (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anaesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202055076
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Penehyclidine; Postoperative Nausea and Vomiting; Bimaxillar Surgery
Keywords: Penehyclidine; Postoperative Nausea and Vomiting; Bimaxillar Surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — penehyclidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): For patients in the control group, a dose of placebo (normal saline 5 ml) is injected intravenously before anesthesia induction. A patient-controlled intravenous analgesia pump is provided after surgery, which is established with a mixture of placebo (normal saline 5 ml), sufentanil (1.25-1.5 ug/kg) and tropisetron 10 mg, diluted with normal saline to 100 ml, and programmed to administer a continuous infusion at a rate of 2 ml/h for 48 hours.
  Interventions: Drug: Placebo
- Single injection group (Experimental): For patients in this group, a dose of penehyclidine (0.5 mg/5 ml) is injected intravenously before anesthesia induction. A patient-controlled intravenous analgesia pump is provided after surgery, which is established with a mixture of placebo (normal saline 5 ml), sufentanil (1.25-1.5 ug/kg) and tropisetron (10 mg), diluted with normal saline to 100 ml, and programmed to administer a continuous infusion at a rate of 2 ml/h for 48 hours.
  Interventions: Drug: Single injection of penehyclidine
- Continuous infusion group (Experimental): For patients in this group, a dose of penehyclidine (0.25 mg/5 ml) is injected intravenously before anesthesia induction. A patient-controlled intravenous analgesia pump is provided after surgery, which is established with a mixture of penehyclidine (0.25 mg/5 ml), sufentanil (1.25-1.5 ug/kg) and tropisetron (10 mg), diluted with normal saline to 100 ml, and programmed to administer a continuous infusion at a rate of 2 ml/h for 48 hours.
  Interventions: Drug: Continuous infusion of penehyclidine

INTERVENTIONS:
Drug: Single injection of penehyclidine — A dose of penehyclidine hydrochloride (0.5 mg/5 ml) is injected intravenously before anesthesia induction. A patient-controlled intravenous analgesia pump is provided after surgery, which is established with a mixture of placebo (normal saline 5 ml), sufentanil (1.25-1.5 ug/kg) and tropisetron (10 mg), diluted with normal saline to 100 ml, and programmed to administer a continuous infusion at a rate of 2 ml/h for 48 hours.
  Other Names: Penehyclidine hydrochloride
  Arms: Single injection group
Drug: Continuous infusion of penehyclidine — A dose of penehyclidine hydrochloride (0.25 mg/5 ml) is injected intravenously before anesthesia induction. A patient-controlled intravenous analgesia pump is provided after surgery, which is established with a mixture of penehyclidine hydrochloride (0.25 mg/5 ml), sufentanil (1.25-1.5 ug/kg) and tropisetron (10 mg), diluted with normal saline to 100 ml, and programmed to administer a continuous infusion at a rate of 2 ml/h for 48 hours.
  Other Names: Penehyclidine hydrochloride
  Arms: Continuous infusion group
Drug: Placebo — A dose of placebo (normal saline 5 ml) is injected intravenously before anesthesia induction. A patient-controlled intravenous analgesia pump is provided after surgery, which is established with a mixture of placebo (normal saline 5 ml), sufentanil (1.25-1.5 ug/kg) and tropisetron (10 mg), diluted with normal saline to 100 ml, and programmed to administer a continuous infusion at a rate of 2 ml/h for 48 hours.
  Other Names: Normal saline
  Arms: Control group

SUMMARY:
Postoperative nausea and vomiting (PONV) is a common complication after surgery. Patients undergoing orthognathic surgery are reported to have a high rate of PONV, especially those undergoing bimaxillary surgery. Activation of cholinergic system plays an important role in the development of PONV. Penehyclidine is an muscarinic antagonists which selectively block M1 and M3 receptors and is commonly used to decrease oral secretion. The investigators hypothesize that continuously administrated penehyclidine during perioperative period can reduce the incidence of PONV in patients undergoing bimaxillary surgery.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is one of the most frequently occurred complications after surgery, and are associated with patients' dissatisfaction after anesthesia and surgery. Orthognathic surgery is widely performed for the correction of dentofacial deformities. Despite of improved anti-emetic prophylaxis, patients undergoing orthognathic surgery are reported to have a high incidence of PONV, especially those after bimaxillary surgery.

It is known that activation of central cholinergic system plays an important role in the development of PONV. Muscarinic antagonists such as scopolamine can block muscarinic receptors in the cerebral cortex and produce anti-emetic effects. Penehyclidine is a new muscarinic antagonists which selectively block M1 and M3 receptors. Our previous study indicated that single-dose of penehyclidine injected before anesthesia induction was associated with a reduced risk of PONV during the first 6 h postoperatively.The mean elimination half-life of penehyclidine following single administration is about 10.35 h. Hence, a single-dose penehyclidine may only produce a short duration of antiemetic effect.

The investigators hypothesize that continuously administrated penehyclidine during perioperative period reduces PONV more effectively than single-dose injection in patients undergoing bimaxillary surgery. The purpose of this study is to investigate the effect of continuous administered penehyclidine in preventing PONV in patients undergoing bimaxillary surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years but <60 years; body mass index ≥18 but <30 kg/m2;
2. Scheduled to undergo elective bimaxillary surgery under general anesthesia;
3. Planned to use patient-controlled intravenous analgesia (PCIA) after surgery;
4. Provide written informed consents.

Exclusion Criteria:

1. Presence of glaucoma;
2. Allergic to penehyclidine, atropine, scopolamine or other anticholinergic drugs;
3. Acute or chronic nausea and/or vomiting, or gastrointestinal motility disorders before surgery;
4. Preoperative antiemetic therapy within 12 hours;
5. History of schizophrenia, Parkinson's disease or profound dementia, or language barrier;
6. Severe hepatic dysfunction (Child-Pugh class C), severe renal dysfunction (requirement of renal replacement therapy before surgery) or American Society of Anesthesiologists physical status ≥IV.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 354 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Incidence of nausea and vomiting within 72 hours after bimaxillary surgery. | Up to 72 hours after surgery.
  Nausea was assessed by direct questioning. Vomiting was diagnosed when patients retched or expulsed intra-gastric contents.

SECONDARY OUTCOMES:
Incidence of nausea and vomiting at different stages after bimaxillary surgery. | Up to 72 hours after surgery.
  Postoperative 0-6 h, 6-12 h, 12-24 h, 24-48 h, and 48-72 h. Nausea was assessed by direct questioning. Vomiting was diagnosed when patients retched or expulsed intra-gastric contents.
Incidence of moderate to severe nausea at different stages after bimaxillary surgery. | Up to 72 hours after surgery.
  Postoperative 0-6 h, 6-12 h, 12-24 h, 24-48 h, and 48-72 h. Severity of nausea is assessed with the numerical rating scale (NRS; an 11-point scale where 0=no nausea and 10=the worst nausea). A score of 4 or higher is defined as moderate to severe nausea.
Incidence of moderate to severe nausea within 72 hours after bimaxillary surgery. | Up to 72 hours after surgery.
  Severity of nausea is assessed with the numerical rating scale (NRS; an 11-point scale where 0=no nausea and 10=the worst nausea). A score of 4 or higher is defined as moderate to severe nausea.
Severity of nausea and vomiting within 72 hours after bimaxillary surgery. | Up to 72 hours after surgery.
  Level I: Absence of any emetic symptoms and nausea during the entire study period.
  Level II: Occurrence of mild nausea or one episode of vomiting if caused by an exogenous stimulus (e.g., drinking or movement).
  Level III: Moderate to severe nausea, or vomiting for 2 times or more, or experiences nausea that required a rescue antiemetic therapy only once.
  Level IV: Patient is suffered more than two emetic episodes or necessitating more than one dose of a rescue antiemetic.
Use of rescue antiemetics within 72 hours after bimaxillary surgery. | Up to 72 hours after surgery.
  Frequency and dose of antiemetics.
Incidence of delirium within the first 5 days after surgery | Up to 5 days after surgery.
  Incidence of delirium within the first 5 days after surgery.
Length of stay in hospital after surgery. | Up to 30 days after surgery.
  Length of stay in hospital after surgery.
Incidence of complications within 30 days after surgery. | Up to 30 days after surgery.
  Incidence of complications within 30 days after surgery.
All-cause 30-day mortality. | Within 30 days after surgery.
  All-cause 30-day mortality.
Cognitive function on the 30th day after surgery. | At 30 days after surgery
  Cognitive function is assessed with the modified Telephone Interview for Cognitive Status (TICS-m; a 12-item questionnaire that provides an assessment of global cognitive function by verbal communication via telephone. The score ranges from 0 to 50, with higher score indicating better function).

OTHER OUTCOMES:
Incidence of moderate to severe pain at different stages after bimaxillary surgery. | Up to 72 hours after surgery.
  Postoperative 0-6 h, 6-12 h, 12-24 h, 24-48 h, and 48-72 h. Pain intensity is assessed with the numerical rating scale (NRS; an 11-point scale where 0=no pain and 10=the worst pain). A score of 4 or higher is defined as moderate to severe pain.
Use of rescue analgesics within 72 hours after bimaxillary surgery. | Up to 72 hours after surgery.
  Frequency and dose of analgesics.
Subjective sleep quality within 3 days after bimaxillary surgery. | In the morning of the 1st, 2nd, and 3rd days after surgery.
  Subjective sleep quality is assessed with the numeric rating scale (NRS; an 11-point scale where 0=the worst sleep and 10=the best sleep).

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking Univeristy Hospital Stomatology, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Myles PS, Williams DL, Hendrata M, Anderson H, Weeks AM. Patient satisfaction after anaesthesia and surgery: results of a prospective survey of 10,811 patients. Br J Anaesth. 2000 Jan;84(1):6-10. doi: 10.1093/oxfordjournals.bja.a013383. PMID 10740539
- [Background] Naran S, Steinbacher DM, Taylor JA. Current Concepts in Orthognathic Surgery. Plast Reconstr Surg. 2018 Jun;141(6):925e-936e. doi: 10.1097/PRS.0000000000004438. PMID 29794714
- [Background] Laskin DM, Carrico CK, Wood J. Predicting postoperative nausea and vomiting in patients undergoing oral and maxillofacial surgery. Int J Oral Maxillofac Surg. 2020 Jan;49(1):22-27. doi: 10.1016/j.ijom.2019.06.016. Epub 2019 Jun 21. PMID 31230771
- [Background] Phillips C, Brookes CD, Rich J, Arbon J, Turvey TA. Postoperative nausea and vomiting following orthognathic surgery. Int J Oral Maxillofac Surg. 2015 Jun;44(6):745-51. doi: 10.1016/j.ijom.2015.01.006. Epub 2015 Feb 2. PMID 25655765
- [Background] Dobbeleir M, De Coster J, Coucke W, Politis C. Postoperative nausea and vomiting after oral and maxillofacial surgery: a prospective study. Int J Oral Maxillofac Surg. 2018 Jun;47(6):721-725. doi: 10.1016/j.ijom.2017.11.018. Epub 2018 Jan 1. PMID 29301675
- [Background] Shaikh SI, Nagarekha D, Hegade G, Marutheesh M. Postoperative nausea and vomiting: A simple yet complex problem. Anesth Essays Res. 2016 Sep-Dec;10(3):388-396. doi: 10.4103/0259-1162.179310. PMID 27746521
- [Background] Han XY, Liu H, Liu CH, Wu B, Chen LF, Zhong BH, Liu KL. Synthesis of the optical isomers of a new anticholinergic drug, penehyclidine hydrochloride (8018). Bioorg Med Chem Lett. 2005 Apr 15;15(8):1979-82. doi: 10.1016/j.bmcl.2005.02.071. PMID 15808451
- [Background] Zhang Z, Zhuang Y, Ouyang F, Zhang A, Zeng B, Gu M. Penehyclidine enhances the efficacy of tropisetron in prevention of PONV following gynecological laparoscopic surgery. J Anesth. 2012 Dec;26(6):864-9. doi: 10.1007/s00540-012-1443-1. Epub 2012 Aug 10. PMID 22878869
- [Derived] Wang LK, Cheng T, Yang XD, Xiong GL, Li N, Wang DX. Penehyclidine for prevention of postoperative nausea and vomiting following bimaxillary orthognathic surgery: a randomized, double-blind, controlled trial. J Anesth. 2022 Feb;36(1):122-136. doi: 10.1007/s00540-021-03017-4. Epub 2021 Nov 5. PMID 34738161